CLINICAL TRIAL: NCT03743896
Title: An Open Label, Single Dose, Bioavailability Study of Topical Transdermal Glucosamine Cream on the Synovial Fluid Tapped From Osteoarthritic Adult, Male and Female Human Subjects Already Undergoing Arthrocentesis
Brief Title: Transdermal Delivery of Glucosamine to the Synovial Fluid of Male and Female With Knee Osteoarthritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lynk Biotechnologies Pte Ltd (Industry)
Collaborators: T&T Family Health Clinic and Surgery, Singapore (Unknown); Temasek Polytechnic School of Applied Science, Singapore (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: ASC/CPROJ/14/15/16; CTC1600169 (Registry Identifier: Health Sciences Authority Singapore)
Record Dates: First submitted 2018-11-13; First posted 2018-11-16 (Actual); Last update posted 2018-11-16 (Actual); Status verified 2018-11

CONDITIONS: Osteoarthritis, Knee
Keywords: Transdermal Delivery; Glucosamine; Synovial Fluid; Osteoarthritis; Knee; Human; Arthrocentesis
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Protein Glutamine gamma Glutamyltransferase 2; Capsaicin

STUDY DESIGN:
Intervention Model Description: Subjects who agreed to participate in the study could decide to be part of the Control group (no intervention) or the Test group (single dose, topical application of Transdermal Glucosamine Cream)
Masking Description: There is no possibility of subjective bias or placebo effect since the primary outcome is the drug concentration in the synovial fluid. Hence no blinding or randomization needed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): No intervention
- Test group (Experimental): single dose (2g), topical application of Transdermal Glucosamine Cream (containing 10% w/w of glucosamine sulfate)
  Interventions: Drug: Transdermal Glucosamine Cream

INTERVENTIONS:
Drug: Transdermal Glucosamine Cream
  Other Names: TGC® Plus Capsaicin
  Arms: Test group

SUMMARY:
Glucosamine is commonly used as a treatment for Osteoarthritis (OA). While oral administration remains the most commonly used route, topical administration could offer numerous advantages such as targeted delivery to affected joints and overcoming the negative effects of the passage of the drug through the digestive system. The objective of this study is to assess the bioavailability of glucosamine in the synovial fluid of osteoarthritic joints, following the topical application of a commercially available transdermal glucosamine cream. Joint fluid samples will be collected from 2 groups of participants with knee OA: the Control group will not be subjected to any treatment while the Test group will apply 2g of transdermal glucosamine cream 1 to 3 hours before the joint fluid collection. Glucosamine concentration will be determined and the results obtained from both groups will be compared. This trial will potentially provide data to support that glucosamine can cross the skin and be delivered to the affected joint fluid when formulated in a transdermal cream base.

ELIGIBILITY:
Inclusion Criteria:

* Male and non-pregnant female human subjects
* 21 to 80 years old
* Subjects who need to undergo arthrocentesis (prescribed during prior medical assessment)
* Willingness to follow the protocol requirements

Exclusion Criteria:

* Known allergy to shellfish
* Known history of hypersensitivity to Glucosamine or related drugs.
* Known history of hypersensitivity to Capsaicin (Capsicum extract)
* Known history of skin sensitivity
* Subjects who have taken any kind of glucosamine during the last 24 hours
* Subjects who have taken any kind of treatment for joint pain during the last 24 hours
* Subjects having scars/cut/dermatological abnormality at application site
* Pregnant or nursing women

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2016-05-18 (Actual); Primary Completion 2017-03-10 (Actual); Study Completion 2017-03-10 (Actual)

PRIMARY OUTCOMES:
Concentration of glucosamine in synovial fluid | 1 to 3 hours post-intervention
  For the Test group
Concentration of glucosamine in synovial fluid | At baseline
  For the Control group

CONTACTS AND LOCATIONS:
Overall Officials: Choon Meng Ting, MD, Principal Investigator — T&T Family Health Clinic and Surgery, Singapore
Locations (1):
- T&T Family Heath Clinic and Surgery, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-21): https://cdn.clinicaltrials.gov/large-docs/96/NCT03743896/Prot_SAP_000.pdf